CLINICAL TRIAL: NCT01791816
Title: Mechanisms of Vasovagal Syncope
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Julian Stewart, Professor of Pediatrics, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1R01HL112736-01A1 (NIH)
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Vasovagal Syncope; Postural Tachycardia Syndrome
Keywords: Vasovagal Syncope; Postural Tachycardia Syndrome; Orthostatic Intolerance; Nitric Oxide (NO); Orthostatic Stress; L-Ng-monomethyl Arginine (L-NMMA); Phenylephrine; Sodium Nitroprusside
MeSH Terms: conditions — Syncope, Vasovagal; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance | interventions — Phenylephrine; omega-N-Methylarginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phenylephrine and L-Ng-monomethyl Arginine (L-NMMA) (Experimental)
  Interventions: Drug: Phenylephrine; Drug: L-Ng-monomethyl Arginine (L-NMMA)

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine dose-response comprises infusion of 0.5, 1, 2, 3, 4 micrograms/kg/min for 10 min at each dose.
  If bloods pressure increases by 30% or if heart rate decreases below 40 beats per minute we will stop infusion.
Drug: L-Ng-monomethyl Arginine (L-NMMA) — Systemic L-NMMA is infused as a 500μg/kg/min loading dose for 15 min followed by a 50μg/kg/min maintenance dose for the remainder of the experiment.

SUMMARY:
Vasovagal Syncope (simple postural faint) is the most common cause of acute loss of consciousness. Postural tachycardia syndrome(POTS) is the most common chronic form of postural lightheadedness. Together they afflict many Americans, mostly young women, who are prevented from gainful employ or school attendance. The underlying mechanism is not known. Our past work suggests that a simple molecule, nitric oxide, acts to subvert normal blood flow controls causing blood to pool in the gut when standing. Our proposal will show the mechanism behind this problem and will indicate effective medical treatments. Patients will be compared to healthy control subjects.

DETAILED DESCRIPTION:
Vasovagal Syncope (VVS,simple faint) is the most common cause of transient loss of consciousness and is the acute episodic form of orthostatic intolerance(OI). Postural tachycardia syndrome (POTS) is the common chronic form of OI. Both are defined by debilitating symptoms and signs while upright relieved by recumbency. Pathophysiological mechanisms have remained elusive although our past work shows that excessive upright central hypovolemia results from splanchnic pooling due to defective splanchnic arterial and venous constriction. Preliminary data support the hypothesis that production of nitric oxide (NO) is enhanced in these patients resulting in reduced sympathetic noradrenergic neurotransmission at pre-junctional and post-junctional sites. Our approach is two-fold: 1) We will use intradermal microdialysis and laser Doppler flowmetry (LDF) to delineate the microvascular mechanisms of NO modulation of noradrenergic neurotransmission free of confounding systemic reflex changes. 2) We will systemically apply this mechanism to a model of orthostatic stress, lower body negative pressure(LBNP), while measuring cardiac output by inert gas rebreathing, regional blood volume, and regional blood flow using plethysmographic techniques focusing on splanchnic changes, and muscle sympathetic nerve activity by peroneal microneurography. We will study synaptic peripheral neurotransmission of Norepinephrine and how it is affected by supplemental NO and by nitric oxide synthase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. POTS patients referred for day to day orthostatic intolerance with greater than 3 symptoms for greater than 3 months and will have the diagnosis of symptomatic postural tachycardia made during a screening tilt table test :

   * dizziness
   * nausea and vomiting
   * palpitations
   * fatigue
   * headache
   * exercise intolerance
   * blurred vision
   * abnormal sweating heat.
2. Vasovagal Syncope patients will have at least 3 episodes of fainting episodes in the past year.
3. Healthy control subjects

Cases will be between the ages of 14 and 29 years old Cases will have normal physical examination, and normal electrocardiographic and echocardiographic evaluations.

Only those free from heart disease, and from systemic illness will be eligible to participate.

This excludes patients with illnesses and disease states known to be associated with endothelial cell dysfunction such as diabetes, renal disease, congestive heart failure, systemic hypertension, acute and chronic inflammatory diseases, neoplasm, immune mediated disease, trauma, morbid obesity and peripheral vascular disease.

At the time of testing all patients and control subjects must refrain from vasoactive drugs for two weeks. Please check with us about any medication that you are taking.

Exclusion Criteria:

* Cardiovascular causes of syncope
* An active medical condition that may explain the diagnosis
* A previous medical condition with undocumented resolution that may explain the diagnosis
* Past or present major psychiatric disorder
* Substance abuse within 2 years before onset of symptoms.

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-02; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Heart rate and blood pressure in response to Lower Body Negative Pressure(LBNP) | 1 year

SECONDARY OUTCOMES:
Adrenergic neurotransmission as measured by Muscle Sympathetic Nerve Activity(MSNA), doppler ultrasound blood flow, venous Norepinephrine in response to Phenylephrine infusion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julian M. Stewart, M.D., Ph.D., Principal Investigator — New York Medical College
Locations (1):
- New York Medical College/Bradhurst Building, Hawthorne, New York, United States

REFERENCES:
- See also: The Center for Hypotension — http://syncope.org/